CLINICAL TRIAL: NCT03634761
Title: Early Intervention and Autism: Transformation From Research to Practice Through a Competency Based Model
Acronym: AUT-TID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lise Roll-Pettersson, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VR 2015-01212
Record Dates: First submitted 2018-05-30; First posted 2018-08-16 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Program Quality; Intervention Setting; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: The study used a staggered design where three waves of preschools were recruited and assigned to either the experimental or the control group. The first wave of preschools (n = 6) were divided into two groups, where group assignment was made to make the two groups comparable in regards to three variables: supervisors' experience of comprehensive programs, APERS-P-SE baseline scores, and children's adaptive behavior (Vineland II ratings). Originally, the plan was to then randomize which of these two matched groups would be the experimental group, but because of unforeseen circumstances one of the groups was made the control group because there was a lack of resources for one of the preschools to be able to be in the experimental group. However, for the following two waves of recruitment, the participating preschools (n = 11) were divided into matched pairs (based only on supervisor experience), which were then randomly assigned either as the control or the experimental group.
Masking Description: In total, 17 preschools, 17 children (one from each preschool), and 35 preschool staff (two from each preschool except from one preschool where three preschool staff participated) participated in the study. None of the participants were blind to their assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Preschools/Children in this group will receive EIBI supervised by an external expert from the habilitation center on a regular basis. In addition, preschool staff in this group are provided with in-service training consisting of a one full day (onset of project) and a half day (middle of project) on autism, applied behavior analysis, evidence-based practices, engagement, participation, inclusion and overall quality factors when working with Children with autism in preschool settings. Preschool staff are also provided with monthly on-site coaching in implementing evidence based practices, goal setting and working with overall intervention setting, through coaching from the habilitation center.
  Interventions: Behavioral: Competency based model; Behavioral: Comprehensive program
- Comparison group (Active Comparator): Preschools/Children are in this group receive "treatment as usual", which is EIBI supervised by an external expert from the habilitation center at the habilitation center directed toward the paraprofessional. At the offset of the project preschool staff are offered to participate in a one-day learning course/workshop on autism, applied behavior analysis, evidence-based practices, engagement, participation, inclusion and overall quality factors when working with children with autism in preschool settings.
  Interventions: Behavioral: Comprehensive program

INTERVENTIONS:
Behavioral: Competency based model — Qualified Learning course and workshop to preschool staff combined with monthly on-site coaching at preschool sites to improve overall intervention setting quality and use of evidence bases practices, provided by external expert from habilitation center.
  Arms: Experimental group
Behavioral: Comprehensive program — Comprehensive program of EIBI for Children with ASD supervised by external expert from habilitation center (treatment as usual)

SUMMARY:
This study evaluates the effect of a competency based model on program quality in Swedish preschools for Children with autism spectrum disorder (ASD). Half of the participating preschools will receive "treatment as usual" (Early Intensive Behavioral Intervention (EIBI) provided to a Child with ASD in the preschool, supervised by an external supervisor from a habilitation center), while the other half will receive the above as well as, in-service training and monthly on-site coaching sessions also involving preschool staff other than the paraprofessional (competency based model). It is hypothesized that the competency based model will improve program quality, child's engagement, preschool staff knowledge, allegiance and self-efficacy compared to the comparison group.

DETAILED DESCRIPTION:
Almost all children in Sweden between two and five years attend preschool including children with Autism spectrum disorder (ASD). High quality and structured early intervention programs grounded in the principles and procedures of applied behavior analysis have been found in numerous research studies and reviews to significantly improve developmental outcomes, adaptive behaviors and learning outcomes of preschool children with ASD.

A prerequisite of which is a high quality learning environment that includes both the physical set-up, learning climate and competence of staff. The primary purpose of this project is to improve program quality for preschool children with ASD through a competency based model grounded in ecological systems theory sustainable over time and applicable within the Swedish service support system. In total approximately 16 preschools will participate, half of which will receive "treatment as usual" EIBI to a Child with ASD in the preschool, supervised by an external supervisor from a habilitation center), while the other half will also receive obtain in-service training and monthly on-site coaching through habilitation. Involved habilitation specialists will obtain in-service training prior to the onset of the study on how to use the Autism Program Environment Rating Scale (APERS), the basic tenets of coaching based on the concept of reflective and collaborative dialogues in which the preschool teachers knowledge of the child and context are taken into account.

It is hypothesized that the competency based model will improve program quality, child's engagement, adaptive behavior, increase preschool staff knowledge, allegiance and self-efficacy compared to the comparison group only receiving supervision in implementing a comprehensive program.

ELIGIBILITY:
Inclusion Criteria:

* Autism diagnosis
* Receiving comprehensive program/EIBI implemented in preschool setting with supervision from habilitation center

Exclusion Criteria:

-

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in overall program quality measured by the Autism Program Environment Rating Scale (APERS-P-SE) | Baseline and follow-up (about 9 months from baseline)
  The APERS-P-SE is a rating scale designed to examine the preschool teaching environment of children with ASD in Sweden. It is used to assess overall intervention setting quality over 10 domains including areas such as Personal Independence and Functional Behavior. It consists of 56 items rated on a 5 Point Likert-scale (1= low quality - 5 = high quality) resulting in individual item scores, subdomain scores, domain scores and a total score.

SECONDARY OUTCOMES:
Ethics, Values and Allegiance (EVA) | Baseline and follow-up (about 9 months from baseline)
  A questionnaire used to assess attitude and allegiance to EIBI among preschool staff. 11 items/statements rated on a five point scale (I don't agree at all, to I highly agree)
Evidence Based Practices (EBP) | Baseline and follow-up (about 9 months from baseline)
  A questionnaire designed to assess knowledge, use and implementation skills of evidence based practices for Children with autism among preschool staff. 15 items rated on a 4 point Likert-scale (0 = no knowledge, 3 = high knowledge)
Autism Knowledge Questionnaire (AKQ) | Baseline and follow-up (about 9 months from baseline)
  A questionnaire designed to assess knowledge on ASD among preschool staff. 18 items/statements about autism, answered either yes/no/I dont know
Self-Efficacy and Stress Questionnaire (SESQ) | Baseline and follow-up (about 9 months from baseline)
  A questionnaire designed to assess stress and self-efficacy among preschool staff working with children with autism. A total of 34 items/statements rated on a 6 point Likert-scale (0 = i don't agree at all, 5 = i fully agree)
Goal Attainment Scale (GAS) | Follow-up about 9 months after onset of study
  An ordinal scale designed to assess level of goal attainment for participating Children in the study rated from 0 (baseline), 1 (initial objective), 2 (secondary objective), 3 (annual goal), 4 (exceeds annual goal)
Clinical Global Impression-autism (CGI-AUT) | Baseline and follow-up (about 9 months from baseline)
  An instrument designed to assess the symptom severity of preschool aged children with ASD rated on a scale between 1 and 7 (1 = no autism symptoms, 7 = maximum symptom severity)
Children's Engagement Questionnaire (CEQ) | Baseline and follow-up (about 9 months from baseline)
  A scale designed to assess children's level of engagement in various situations in and outside the preschool. It consists of 31 items/situations, rated on a 4 point scale (not at all typical, to very typical)
Vineland Adaptive Behavior Scales - Second Edition (Vineland-II) - Teacher ratings | Baseline and follow-up (about 9 months from baseline)
  A scale designed to assess the adaptive functioning for children within various domains such as independence and Communication skills. Rated on a 3 point scale (0 = never occurs, 2 = occurs often)

OTHER OUTCOMES:
Social validity scale | Follow-up about 9 months after onset of study
  A scale designed to asses the social validity of the goals targeted within the study

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - BanyanCenter, Stockholm
  - Autismcenter för Små Barn, Stockholm